CLINICAL TRIAL: NCT03905070
Title: Investigation of Body Awareness and Affecting Factors in Bariatric Surgery Patients
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ümit VARLI, Principal Investigator, Izmir Katip Celebi University
Other Study IDs: 103
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery; Body Image
Keywords: bariatric surgery; body awareness; physical therapy; metabolic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study Group: The study group consisted of people who had undergone bariatric surgery and who had at least 6 months after the operation.
- Control Group: The control group will consist of asymptomatic individuals whose BMI is 18-25 kg / m2 and has not participated in any exercise program in the last one year.

SUMMARY:
The aim of this study is to investigate the body awareness and the factors affecting the bariatric surgery.

DETAILED DESCRIPTION:
In the treatment of obesity, bariatric surgery allows for significant and permanent weight loss and is the most effective treatment. Although the effect of changing body image on occupational and social experiences in patients undergoing bariatric surgery has been examined, there is not enough information about the body awareness and the factors affecting these patients. The aim of this study is to investigate the body awareness and the factors affecting the bariatric surgery.

In this study, body composition (with body analyzer), body awareness (with Body Awareness Questionnaire), physical activity level (with International Physical Activity Questionnaire-Short Form), joint position feeling (with photography method), quality of life (with Short Form-36), depression status (with Beck Depression Inventory) and cognition (with Montreal Cognitive Assessment Test) of all participants will be evaluated when they come routine doctor control.

ELIGIBILITY:
Inclusion Criteria:

* Having a bariatric surgery,
* At least 6 months after surgery
* Being between the ages of 18-65,
* To read and understand Turkish
* Volunteer to participate in the study

Exclusion Criteria:

* Musculoskeletal problems to prevent the tests to be applied,
* Psychiatric diagnosis,
* Drinking alcohol and / or drugs,
* Refusal to volunteer

For the control group to be included in the study, the BMI should be between 18-25 kg / m2, read and write in Turkish, and be voluntary. Those who have been included in any exercise program (plates, yoga, dance, etc.) in the last 1 year will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be two groups in the study: Study and Control groups. The study group consisted of people who had undergone bariatric surgery and who had at least 6 months after the operation. The control group will consist of asymptomatic individuals whose BMI is 18-25 kg / m2 and has not participated in any exercise program in the last one year.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Body Awareness | Data collection will continue until September 2019. Data analysis and report preparation will be completed by December 2019.
  Body awareness of patients will be evaluated with Body Awareness Questionnaire (BAQ). It is a survey of 18 statements. Each statement is scored from 1 to 7 points. The total score can be 18 to 126. High score indicates that body awareness is good.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur NAZ GÜRŞAN, PhD, Study Director — Izmir Katip Celebi University, Faculty of Health Science
Locations (1):
- Izmir Katip Celebi University, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the study is completed and published, the investigators are considering the update the plan.

REFERENCES:
- [Background] Morana C, Collignon M, Nocca D. Effectiveness of a Functional Rehabilitation Program After Bariatric Surgery: a Pilot Study. Obes Surg. 2018 Aug;28(8):2321-2326. doi: 10.1007/s11695-018-3154-7. PMID 29484608
- [Background] Major P, Matlok M, Pedziwiatr M, Migaczewski M, Budzynski P, Stanek M, Kisielewski M, Natkaniec M, Budzynski A. Quality of Life After Bariatric Surgery. Obes Surg. 2015 Sep;25(9):1703-10. doi: 10.1007/s11695-015-1601-2. PMID 25676156
- [Background] Mundbjerg LH, Stolberg CR, Cecere S, Bladbjerg EM, Funch-Jensen P, Gram B, Juhl CB. Supervised Physical Training Improves Weight Loss After Roux-en-Y Gastric Bypass Surgery: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 May;26(5):828-837. doi: 10.1002/oby.22143. Epub 2018 Mar 22. PMID 29566463
- [Background] Natvik E, Groven KS, Raheim M, Gjengedal E, Gallagher S. Space perception, movement, and insight: attuning to the space of everyday life after major weight loss. Physiother Theory Pract. 2019 Feb;35(2):101-108. doi: 10.1080/09593985.2018.1441934. Epub 2018 Feb 27. PMID 29485300
- [Background] Skjaerven LH, Mattsson M, Catalan-Matamoros D, Parker A, Gard G, Gyllensten AL. Consensus on core phenomena and statements describing Basic Body Awareness Therapy within the movement awareness domain in physiotherapy. Physiother Theory Pract. 2019 Jan;35(1):80-93. doi: 10.1080/09593985.2018.1434578. Epub 2018 Feb 26. PMID 29482403
- [Background] Guardia D, Metral M, Pigeyre M, Bauwens I, Cottencin O, Luyat M. Body distortions after massive weight loss: lack of updating of the body schema hypothesis. Eat Weight Disord. 2013 Sep;18(3):333-6. doi: 10.1007/s40519-013-0032-0. Epub 2013 Apr 20. PMID 23760908
- [Background] Jung F, Spahlholz J, Hilbert A, Riedel-Heller SG, Luck-Sikorski C. Impact of Weight-Related Discrimination, Body Dissatisfaction and Self-Stigma on the Desire to Weigh Less. Obes Facts. 2017;10(2):139-151. doi: 10.1159/000468154. Epub 2017 Apr 22. PMID 28434008
- [Background] Warholm C, Marie Oien A, Raheim M. The ambivalence of losing weight after bariatric surgery. Int J Qual Stud Health Well-being. 2014 Jan 29;9:22876. doi: 10.3402/qhw.v9.22876. eCollection 2014. PMID 24480033